CLINICAL TRIAL: NCT07271771
Title: The Effect of Denosumab on Muscle and Strength and Insulin Sensitivity
Acronym: DENMUSIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Sponsor: MD, Professor, DMSc, PhD Bente Lomholt Langdahl (Unknown)
Responsible Party: Principal Investigator, Anne Sophie Sølling, MD, PhD, postdoc, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTIS: 2024-510637-18-00; CTIS: 2024-510637-18-00 (Other: Aarhus University Hospital, Denmark)
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Osteoporosis
Keywords: muscle; insulin sensitivity; denosumab; bone mineral density
MeSH Terms: conditions — Osteoporosis; Insulin Resistance | interventions — Denosumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study is a randomized double-blind, interventional study in 40 postmenopausal with diabetes mellitus type 2. The patients will be randomized at baseline to denosumab 60 mg (n=20) or placebo (n=20), which will administrated at base-line and month 6.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group 1 (Experimental): Denosumab
  Interventions: Drug: Denosumab
- Study group 2 (Placebo Comparator): Placebo
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Denosumab — Denosumab 60 mg
  Arms: Study group 1
Drug: Saline (0.9% NaCl) — Placebo
  Other Names: Placebo
  Arms: Study group 2

SUMMARY:
Randomized, placebo controlled prospective trial evaluating the effect of denosumab on insulin sensitivity and muscle strength.

DETAILED DESCRIPTION:
Denosumab is an antibody against receptor-activator of nuclear factor kappa-B ligand (RANKL) that prevents recruitment and differentiation of mature osteoclasts. Treatment with denosumab markedly decreases bone resorption, increases bone mineral density (BMD), and reduces the risk of vertebral as well as non-vertebral and hip fractures. Osteoclasts produce dipeptidyl peptidase-4 (DPP-4) that degrades glucagon-like peptide-1 (GLP-1) and GLP-1 stimulates insulin production. In accordance with this, animal models have shown a beneficial effect of denosumab on glucose metabolism. However, data from clinical studies in patients with osteoporosis are limited and the results inconsistent. In a small, randomised trial with 52 healthy postmenopausal women, treatment with denosumab for 12 months reduced DPP-4 and increased GLP-1 compared to placebo but no effect was seen on insulin or fasting glucose levels. In the same publication, the authors conducted a non-randomized, observational study in osteoporotic patients with diabetes mellitus or prediabetes that were treated with either denosumab, bisphosphonates, or calcium + vitamin D at the discretion of their physician. Here, treatment with denosumab significantly reduced fasting glucose after 6 months and HbA1c after 12 months compared to bisphosphonates or calcium + vitamin D. Similar findings were seen in another observational study with 20 patients with diabetes. On the other hand, a post hoc analysis of the FREEDOM trial did not find a general effect of denosumab on fasting glucose in postmenopausal women with self-reported diabetes or prediabetes, but only reported a small decrease in fasting glucose in denosumab treated women with diabetes not treated with antidiabetics. This is in line with three small observational studies, in which no clinically relevant effect of denosumab on fasting glucose, insulin level or homeostatic model assessment for insulin resistance (HOMA-IR) was identified.

Overall, the heterogeneity across the studies is large, most of the trials are observational studies and the results are inconsistent. Therefore, randomized, controlled trials are warranted to further elucidate this.

Denosumab has also been shown to improve muscle strength compared to placebo in animal models, however, data from human studies is limited. In an observational study, denosumab decreased the risk of falls and improved sarcopenia measures in 135 patients with osteoporosis compared to 272 patients treated with alendronate or zoledronate assessed at treatment initiation and after 5 years for denosumab and alendronate and 3 years for zoledronate. All outcome measures worsened one years after denosumab discontinuation. In another prospective observational study with 18 postmenopausal women, denosumab treatment for an average of three years improved appendicular lean mass and handgrip strength compared to treatment with bisphosphates or placebo. This is in line with two additional observational studies, in which denosumab improved muscle strength after 6 - 17 months compared to bisphosphonates or vitamin D.

None of the studies evaluating the effect of denosumab on muscle strength are randomised controlled trials, the outcome measures are different and the follow up visits few. Also, none of the studies controlled for exercise.

The investigators therefore want to conduct a randomized, placebo controlled prospective trial evaluating the effect of denosumab on insulin sensitivity and muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (postmenopausal for at least two years)
* Age ≥ 40 years
* BMD T-score ≥ -2.0 (lumbar spine, total hip or femoral neck)
* At least 2 lumbar vertebrae that can be evaluated by dual-energy x-ray absorptiometry (DXA)
* Diabetes Mellitus type 2
* Treatment with metformin as monotherapy

Exclusion Criteria:

* Treatment for osteoporosis at any time
* Other antidiabetic medication than metformin
* Low-energy vertebral fractures at any time
* Low-energy hip fracture at any time
* Ongoing treatment with systemic glucocorticoids
* Metabolic bone disease (for example osteogenesis imperfecta, Paget's disease of bone, hyperparathyroidism)
* Treatment affecting bone, calcium metabolism or muscle
* Active cancer within the last 5 years with the exception of basal cell skin cancer
* Estimated glomerular filtration rate (eGFR) ≤ 35 mL/min
* Unable to read and understand Danish
* Immobility

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity: HbA1c | 12 months
  Changes in Hb1Ac (mmol/mol) from baseline to month 12
Insulin sensitivity: HOMA-IR | 12 months
  Changes in HOMA-IR from baseline to month 12
Insulin sensitivity: fasting glucose | 12 months
  Changes in fasting glucose (mmol/l) from baseline to month 12
Insulin sensitivity: oral glucose tolerance test | 12 months
  Changes in oral glucose tolerance test (OGTT) (mmol/l) from baseline to month 12
Muscle mass | 12 months
  Changes in muscle mass (kg) from baseline to month 12.
Muscle strength | 12 months
  Changes in muscle strength (N) from baseline to month 12.

SECONDARY OUTCOMES:
DPP-4 | 12 months
  Changes in DPP-4 (U/L) from baseline to month 12.
GLP-1 | 12 months
  Changes in GLP-1 (pmol/L) from baseline to month 12.
Bone turnover markers: CTX | 12 months
  Changes in carboxy-terminal collagen crosslinks (CTX) (ug/l) from baseline to month 12.
Bone turnover markers: PINP | 12 months
  Changes in procollagen type I N-terminal propeptide (PINP) (ug/L) from baseline to month 12.
Bone Mineral Density | 12 months
  Change in lumbar spine BMD (g/cm2) from baseline to month 12.
Advanced glycation end products (AGEs) | 12 months
  Change in advanced glycation end products (AGEs) from baseline to month 12.
Muscle strength | Month 1 and 3
  Changes in muscle strength (N) from baseline to month 1 and 3.
Insulin sensitivity: Hb1Ac month 1 and 3 | Month 1 and 3
  Changes in Hb1Ac (mmol/mol) from baseline to month 1 and 3
Insulin sensitivity: HOMA-IR month 1 and 3 | Month 1 and 3
  Changes in HOMA-IR from baseline to month 1 and 3
insulin sensitivity: fasting glucose month 1 and 3 | Month 1 and 3
  Changes in fasting glucose (mmol/l) from baseline to month 1 and 3
Insulin sensitivity: OGTT month 1 and 3 | Month 1 and 3
  Changes in oral glucose tolerance test (OGTT) (mmol/l) from baseline to month 1 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Bente Langdahl, MD, Professor, DMSc, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
All results including inconclusive, positive, and negative results will be accessible to the public after the study has ended. As soon as possible and no later than one year after the trial has ended, the trial results will be submitted to the CTIS-portal.

REFERENCES:
- [Background] Anastasilakis AD, Papapoulos SE, Polyzos SA, Appelman-Dijkstra NM, Makras P. Zoledronate for the Prevention of Bone Loss in Women Discontinuing Denosumab Treatment. A Prospective 2-Year Clinical Trial. J Bone Miner Res. 2019 Dec;34(12):2220-2228. doi: 10.1002/jbmr.3853. Epub 2019 Oct 14. PMID 31433518
- [Background] Miller PD, Bolognese MA, Lewiecki EM, McClung MR, Ding B, Austin M, Liu Y, San Martin J. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone. 2008 Aug;43(2):222-229. doi: 10.1016/j.bone.2008.04.007. Epub 2008 Apr 26. PMID 18539106
- [Background] Rupp T, von Vopelius E, Strahl A, Oheim R, Barvencik F, Amling M, Rolvien T. Beneficial effects of denosumab on muscle performance in patients with low BMD: a retrospective, propensity score-matched study. Osteoporos Int. 2022 Oct;33(10):2177-2184. doi: 10.1007/s00198-022-06470-3. Epub 2022 Jun 25. PMID 35751664
- [Background] Phu S, Bani Hassan E, Vogrin S, Kirk B, Duque G. Effect of Denosumab on Falls, Muscle Strength, and Function in Community-Dwelling Older Adults. J Am Geriatr Soc. 2019 Dec;67(12):2660-2661. doi: 10.1111/jgs.16165. Epub 2019 Sep 4. No abstract available. PMID 31483858
- [Background] Miedany YE, Gaafary ME, Toth M, Hegazi MO, Aroussy NE, Hassan W, Almedany S, Nasr A, Bahlas S, Galal S; Egyptian Academy of Bone Health, Metabolic Bone Diseases. Is there a potential dual effect of denosumab for treatment of osteoporosis and sarcopenia? Clin Rheumatol. 2021 Oct;40(10):4225-4232. doi: 10.1007/s10067-021-05757-w. Epub 2021 May 19. PMID 34008069
- [Background] Rossini A, Frigerio S, Dozio E, Trevisan R, Perseghin G, Corbetta S. Effect of Denosumab on Glucose Homeostasis in Postmenopausal Women with Breast Cancer Treated with Aromatase Inhibitors: A Pilot Study. Int J Endocrinol. 2020 Nov 6;2020:1809150. doi: 10.1155/2020/1809150. eCollection 2020. PMID 33204260
- [Background] Lasco A, Morabito N, Basile G, Atteritano M, Gaudio A, Giorgianni GM, Morini E, Faraci B, Bellone F, Catalano A. Denosumab Inhibition of RANKL and Insulin Resistance in Postmenopausal Women with Osteoporosis. Calcif Tissue Int. 2016 Feb;98(2):123-8. doi: 10.1007/s00223-015-0075-5. Epub 2015 Oct 24. PMID 26498169
- [Background] Passeri E, Benedini S, Costa E, Corbetta S. A Single 60 mg Dose of Denosumab Might Improve Hepatic Insulin Sensitivity in Postmenopausal Nondiabetic Severe Osteoporotic Women. Int J Endocrinol. 2015;2015:352858. doi: 10.1155/2015/352858. Epub 2015 Mar 19. PMID 25873952
- [Background] Napoli N, Pannacciulli N, Vittinghoff E, Crittenden D, Yun J, Wang A, Wagman R, Schwartz AV. Effect of denosumab on fasting glucose in women with diabetes or prediabetes from the FREEDOM trial. Diabetes Metab Res Rev. 2018 May;34(4):e2991. doi: 10.1002/dmrr.2991. Epub 2018 Apr 16. PMID 29430796
- [Background] Abe I, Ochi K, Takashi Y, Yamao Y, Ohishi H, Fujii H, Minezaki M, Sugimoto K, Kudo T, Abe M, Ohnishi Y, Mukoubara S, Kobayashi K. Effect of denosumab, a human monoclonal antibody of receptor activator of nuclear factor kappa-B ligand (RANKL), upon glycemic and metabolic parameters: Effect of denosumab on glycemic parameters. Medicine (Baltimore). 2019 Nov;98(47):e18067. doi: 10.1097/MD.0000000000018067. PMID 31764838
- [Background] Bonnet N, Bourgoin L, Biver E, Douni E, Ferrari S. RANKL inhibition improves muscle strength and insulin sensitivity and restores bone mass. J Clin Invest. 2019 May 23;129(8):3214-3223. doi: 10.1172/JCI125915. PMID 31120440
- [Background] Weivoda MM, Chew CK, Monroe DG, Farr JN, Atkinson EJ, Geske JR, Eckhardt B, Thicke B, Ruan M, Tweed AJ, McCready LK, Rizza RA, Matveyenko A, Kassem M, Andersen TL, Vella A, Drake MT, Clarke BL, Oursler MJ, Khosla S. Identification of osteoclast-osteoblast coupling factors in humans reveals links between bone and energy metabolism. Nat Commun. 2020 Jan 7;11(1):87. doi: 10.1038/s41467-019-14003-6. PMID 31911667
- [Background] Bone HG, Wagman RB, Brandi ML, Brown JP, Chapurlat R, Cummings SR, Czerwinski E, Fahrleitner-Pammer A, Kendler DL, Lippuner K, Reginster JY, Roux C, Malouf J, Bradley MN, Daizadeh NS, Wang A, Dakin P, Pannacciulli N, Dempster DW, Papapoulos S. 10 years of denosumab treatment in postmenopausal women with osteoporosis: results from the phase 3 randomised FREEDOM trial and open-label extension. Lancet Diabetes Endocrinol. 2017 Jul;5(7):513-523. doi: 10.1016/S2213-8587(17)30138-9. Epub 2017 May 22. PMID 28546097
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] Lacey DL, Boyle WJ, Simonet WS, Kostenuik PJ, Dougall WC, Sullivan JK, San Martin J, Dansey R. Bench to bedside: elucidation of the OPG-RANK-RANKL pathway and the development of denosumab. Nat Rev Drug Discov. 2012 May;11(5):401-19. doi: 10.1038/nrd3705. PMID 22543469

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT07271771/Prot_SAP_000.pdf